CLINICAL TRIAL: NCT05876702
Title: Endoscopic I-scan Versus Histopathological Evaluation Of Esophageal Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Michael Mokhtar Sadik, Resident-Tropical medecine department-sohag hospital university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-23-05-05MS
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Esophageal Lesions
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: endoscopy — use of upper endoscopy with i-scan specially , in diagnosis of esophageal lesions and comparison of results with histopathology.

SUMMARY:
Considering esophageal diseases, according to a cross-sectional study of endoscopic findings in patients who underwent upper endoscopy at the Fayoum University Hospital, the most common esophageal conditions seen with the endoscope were esophageal varices (25.6% of cases), GERD (23.8% of cases), esophagitis (7.4% of cases), and esophageal monilasis.

GERD is characterized by dystressing symptoms and consequences brought on by the reflux of stomach contents. (Vakil et al., 2006)It appears that the 2 main GERD phenotypes have different pathophysiological and clinical characteristics. In addition, the response to antireflux medication varied significantly between NERD and erosive esophagitis. Patients with NERD made up the majority of the group with refractory heartburn because they had a noticeably lower response rate to proton pump inhibitor (PPI) therapy.

Barrett's oesophagus (BO) and oesophageal adenocarcinoma, may develop as a result of GERD. Barrett's oesophagus is characterised by intestinal metaplasia, which is characterised by acid mucin-containing goblet cells, and the replacement of any length of the squamous epithelium in the distal oesophagus by columnar epithelium.

Dysphagia is frequently brought on by esophageal cancer, which is a serious public health issue. In 2003, there were an estimated 13,900 new instances of esophageal cancer in the US, and 13,000 people passed away from the disease. Only 13% of people survive five years.

High-resolution white-light endoscopy during gastroscopy can identify abnormalities in the mucosa. The endoscopist must decide if the aetiology of erosions, ulcers, strictures, or metaplasia is non-neoplastic or cancerous if they are discovered. Discoloration, a grainy appearance (orange peel effect), and small lumps and depressions in Barrett's layer are indications of dysplasia.

The high-definition I-Scan was created by Pentax (HOYA, Japan) and is based on processing the picture captured by the endoscope's CCD (charge coupled device) to enhance the contrast of the vascular structures and the patterns of the digestive tract's mucosa.(Andrés Reyes-Dorantes, 2011)For the situations outlined below, some authors advise using the I-Scan modes:I-Scan 1 (SE) thought to be used to find lesions. Without affecting the clarity of the endoscopic image, it sharpens the image of minute surface defects,the I-Scan 2 (TE plus SE) imaging system should be utilized to characterize lesions. It increases subtle alterations in the mucosa and vascular architecture while combining surface and tone augmentation and for defining lesions, I-Scan 3 (TE plus CE) should be utilized. The margins of the endoscopic image are darkened and blue colour is digitally added.

In patients with gastrointestinal diseases, endoscopic biopsy and histological evaluation enable early diagnosis of precancerous and cancerous tumours and prompt disease therapy.(Afzal et al., 2006)The results of specimens from a study conducted over five years (2004-2008) in the pathology departments of Cairo University's faculty of medicine and the Theodor Bilharz Research Institute in Egypt were as follows: 54.76% of the 210 esophageal specimens had GERD, 17.61% had Barrett's oesophagus, 3.81% had benign lesions, 18.6% had malignant lesions (squamous cell carcinoma, adenocarcinoma, and undifferentiated carcinoma, each accounting for 10.48% of the total), and 5.24% had other conditions.

ELIGIBILITY:
Inclusion Criteria:

* : All patients with any gastro-esophageal symptoms who underwent upper endoscopy at the endoscopy unit of Tropical medicine and Gastroenterology department will be included.

Exclusion Criteria:

* Any cirrhotic patient.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
detection of esophageal lesions | 12 months
  comparison between number of lesions that could be detected by upper endoscopy and lesions detected by histopathological examination of taken biopsies

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fass R, Sifrim D. Management of heartburn not responding to proton pump inhibitors. Gut. 2009 Feb;58(2):295-309. doi: 10.1136/gut.2007.145581. PMID 19136523
- [Background] Galloro G. High technology imaging in digestive endoscopy. World J Gastrointest Endosc. 2012 Feb 16;4(2):22-7. doi: 10.4253/wjge.v4.i2.22. PMID 22347528
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2019. CA Cancer J Clin. 2019 Jan;69(1):7-34. doi: 10.3322/caac.21551. Epub 2019 Jan 8. PMID 30620402
- [Background] Spechler SJ. Barrett esophagus and risk of esophageal cancer: a clinical review. JAMA. 2013 Aug 14;310(6):627-36. doi: 10.1001/jama.2013.226450. PMID 23942681
- [Background] Vakil N, van Zanten SV, Kahrilas P, Dent J, Jones R; Global Consensus Group. The Montreal definition and classification of gastroesophageal reflux disease: a global evidence-based consensus. Am J Gastroenterol. 2006 Aug;101(8):1900-20; quiz 1943. doi: 10.1111/j.1572-0241.2006.00630.x. PMID 16928254